CLINICAL TRIAL: NCT00810303
Title: Pharmacokinetic and Pharmacodynamic Interactions Between the Cholesterol-lowering Ezetimibe and the Non-nucleoside Reverse Transcriptase Inhibitor Efavirenz During Chronic Treatment in Healthy Volunteers With Reference to Intestinal Expression of CYP3A4, UGT1A1, ABCB1 and ABCC2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Prof. Dr. W. Siegmund, MD, Organization: Department of Clinical Pharmacology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Efavirenz - 2008
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-09

CONDITIONS: Pharmacokinetics; Drug Interactions; Pharmacodynamics; Intestinal Transporter Expression
MeSH Terms: interventions — Ezetimibe; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- whole study group (Experimental): A study with a duration of 34 days with 4 periods (= 4 pharmakokinetics) on 12 healthy subjects.
  Interventions: Drug: Ezetrol (ezetimibe) multiple dose; Drug: Ezetrol (ezetimibe) multiple dose and Sustiva (efavirenz) single dose; Drug: Ezetrol (ezetimibe) and Sustiva (efavirenz) multiple dose; Drug: Sustiva (efavirenz) single dose

INTERVENTIONS:
Drug: Ezetrol (ezetimibe) multiple dose — administration of 1 tablet/day Ezetrol (10 mg ezetimibe) on study day 6-15 and a pharmakokinetic on study day 15 (0-24 h blood sampling, 0-24 h urine sampling and 5 d feces sampling (study day 11-15))
  Other Names: Ezetrol
Drug: Ezetrol (ezetimibe) multiple dose and Sustiva (efavirenz) single dose — administration of 1 tablet/day Ezetrol(R) (10 mg ezetimibe) on study day 16-20 and 2 capsules Sustiva(R) (2x200 mg efavirenz) on study day 16 with a pharmakokinetic (0-120 h blood sampling, urine sampling (24 h intervals) and feces sampling on study days 16-20)
  Other Names: Ezetrol+Sustiva single dose
Drug: Ezetrol (ezetimibe) and Sustiva (efavirenz) multiple dose — administration of 1 tablet/day Ezetrol(R) (10 mg ezetimibe) and 2 capsules/day Sustiva(R) (2x200 mg efavirenz) on study day 21-30 and with a pharmakokinetic (0-120 h blood sampling, urine sampling (24 h intervals) on study day 30 and feces sampling on study day 26-30)
  Other Names: Ezetrol+Sustiva steady state
Drug: Sustiva (efavirenz) single dose — administration of 2 capsules Sustiva(R) (2x200 mg efavirenz) on study day 1 with a pharmakokinetic (0-120 h blood sampling, urine sampling (24 h intervals) and feces sampling on study days 1-5)
  Other Names: Sustiva

SUMMARY:
The purpose of this study is to evaluate the effects of a chronic co-medication of efavirenz on pharmacokinetics and sterol-lowering effects of ezetimibe at steady-state in healthy subjects genotyped for ABCB1, ABCC2, CYP2B6 and UGT1A1.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: Caucasian
* body weight: 19 to 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* existing cardiac or haematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* existing hepatic and renal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* existing gastrointestinal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* acute or chronic diseases which could affect drug absorption or metabolism
* history of any serious psychological disorder
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive anti-HIV-test, HBs-Ag-test or anti-HCV-test
* volunteers who are on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* lactation and pregnancy test positive or not performed
* volunteers suspected or known not to follow instructions
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* volunteers liable to orthostatic dysregulation, fainting, or blackouts
* blood donation or other blood loss of more than 400 ml within the last 12 weeks prior to the start of the study
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* any systemically available medication within 4 weeks prior to the intended first administration unless because of the terminal elimination half-life complete elimination from the body can be assumed for the drug and/or its primary metabolites (except oral contraceptives)
* repeated use of drugs during the last 4 weeks prior to the intended first administration, which can influence hepatic biotransformation (e.g. barbiturates, cimetidine, phenytoin, rifampicin)
* repeated use of drugs during the last 2 weeks prior to the intended first administration which affect absorption (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists)
* intake of grapefruit containing food or beverages within 7 days prior to administration
* known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparation
* subjects with severe allergies or multiple drug allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Greifswald, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: whole study group: 12 healthy subjects
Period: Efavirenz Alone - Day 1-5
Arm/Group | Study Group
Started | 12
Completed | 12
Not Completed | 0
Period: Ezetimibe Alone - Day 6-15
Arm/Group | Study Group
Started | 12
Completed | 12
Not Completed | 0
Period: Ezetimibe and Efavirenz - Day 16-20
Arm/Group | Study Group
Started | 12
Completed | 12
Not Completed | 0
Period: Ezetimibe and Efavirenz - Day 21-30
Arm/Group | Study Group
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  Germany | 12

OUTCOME MEASURES:

1. Primary Outcome: AUC0-24h of Free Ezetimibe (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe) on Study Day 15
Description: The area under the concentrations-time curve (AUC0-24) was calculated with the measured data points from the time of administration up to 24 h after administration by the trapezoidal formula. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free ezetimibe in the blood samplings.
Time Frame: study day 15
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 51.9 (21.7)

2. Primary Outcome: AUC0-24h of Free Ezetimibe (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Single Dose Administration of 400 mg Efavirenz) on Study Day 16
Description: as for outcome 1
Time Frame: study day 16
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 58.6 (23.7)

3. Primary Outcome: AUC0-24h of Free Ezetimibe (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Chronic Treatment With 400 mg Efavirenz) on Study Day 30
Description: as for outcome 1
Time Frame: study day 30
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 51.2 (23.1)

4. Primary Outcome: Cmax of Free Ezetimibe (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe) on Study Day 15
Description: The maximum concentration (Cmax) were obtained directly from the measured concentration-time curves. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free ezetimibe in the blood samplings.
Time Frame: study day 15
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 4.82 (2.74)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe alone and free ezetimibe with single dose treatment of efavirenz; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Cmax of Free Ezetimibe (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Single Dose Administration of 400 mg Efavirenz) on Study Day 16
Description: as for outcome 4
Time Frame: study day 16
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 5.54 (2.65)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe alone and free ezetimibe with single dose treatment of efavirenz; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Cmax of Free Ezetimibe (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Chronic Treatment With 400 mg Efavirenz) on Study Day 30
Description: as for outcome 4
Time Frame: study day 30
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 4.46 (2.07)

7. Primary Outcome: AUC of Efavirenz (Single Dose Pharmacokinetic After Treatment With 400 mg Efavirenz) on Study Days 1-5
Description: The area under the concentrations-time curve (AUC) was calculated with the measured data points from the time of administration until the last quantificable concentration by the trapezoidal formula and the extrapolation to infinity. The concentration-time curve is the result of time points of blood sampling and its measured concentration of efavirenz in the blood samplings.
Time Frame: study days 1-5
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 29.7 (15.4)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between steady state pharmakokinetic of efavirenz with chronic treatment of ezetimibe and the single dose pharmakokinetic of efavirenz without chronic treatment of ezetimibe; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

8. Primary Outcome: AUC of Efavirenz (Single Dose Pharmacokinetic After Treatment With 400 mg Efavirenz and Concomitant Chronic Treatment of 10 mg Ezetimibe) on Study Days 16-20
Description: as for outcome 7
Time Frame: study days 16-20
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 27.0 (12.2)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between steady state pharmakokinetic of efavirenz with chronic treatment of ezetimibe and the single dose pharmakokinetic of efavirenz with chronic treatment of ezetimibe; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

9. Primary Outcome: AUC0-24h of Efavirenz (Steady State Pharmacokinetic After Chronic Treatment With 400 mg Efavirenz and Concomitant Chronic Treatment of 10 mg Ezetimibe) on Study Day 30
Description: The area under the concentrations-time curve (AUC0-24) was calculated with the measured data points from the time of administration up to 24 h after administration by the trapezoidal formula. The concentration-time curve is the result of time points of blood sampling and its measured concentration of efavirenz in the blood samplings.
Time Frame: study day 30
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 11.4 (4.64)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Group; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Cmax of Efavirenz (Single Dose Pharmacokinetic After Treatment With 400 mg Efavirenz) on Study Days 1-5
Description: The maximum concentration (Cmax) were obtained directly from the measured concentration-time curves. The concentration-time curve is the result of time points of blood sampling and its measured concentration of efavirenz in the blood samplings.
Time Frame: study days 1-5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 0.622 (0.244)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

11. Primary Outcome: Cmax of Efavirenz (Single Dose Pharmacokinetic After Treatment With 400 mg Efavirenz and Concomitant Chronic Treatment of 10 mg Ezetimibe) on Study Days 16-20
Description: as for outcome 10
Time Frame: study days 16-20
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 0.659 (0.395)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between steady state pharmakokinetic of efavirenz with chronic treatment of ezetimibe and the single dose pharmakokinetics of efavirenz with chronic treatment of ezetimibe; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Cmax of Efavirenz (Steady State Pharmacokinetic After Chronic Treatment With 400 mg Efavirenz and Concomitant Chronic Treatment of 10 mg Ezetimibe) on Study Day 30
Description: as for outcome 10
Time Frame: study day 30
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 0.918 (0.342)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: AUC0-24h of Ezetimibe Glucuronide (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe) on Study Day 15
Description: The area under the concentrations-time curve (AUC0-24) was calculated with the measured data points from the time of administration up to 24 h after administration by the trapezoidal formula. The concentration-time curve is the result of time points of blood sampling and its measured concentration of ezetimibe glucuronide in the blood samplings.
Time Frame: study day 15
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 466 (223)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe alone and free ezetimibe with single dose treatment of efavirenz; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe with chronic treatment of efavirenz and free ezetimibe alone; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: AUC0-24h of Ezetimibe Glucuronide (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Single Dose Administration of 400 mg Efavirenz) on Study Day 16
Description: as for outcome 13
Time Frame: study day 16
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 411 (195)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe alone and free ezetimibe with single dose treatment of efavirenz; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe with chronic treatment of efavirenz and free ezetimibe with single dose treatment of efavirenz; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: AUC0-24h of Ezetimibe Glucuronide (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Chronic Treatment With 400 mg Efavirenz) on Study Day 30
Description: as for outcome 13
Time Frame: study day 30
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng*h/ml | 325 (152)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe with chronic treatment of efavirenz and free ezetimibe alone; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Group; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Cmax of Ezetimibe Glucuronide (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe) on Study Day 15
Description: The maximum concentration (Cmax) were obtained directly from the measured concentration-time curves. The concentration-time curve is the result of time points of blood sampling and its measured concentration of ezetimibe glucuronide in the blood samplings.
Time Frame: study day 15
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 79.0 (43.1)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe with chronic treatment of efavirenz and free ezetimibe alone; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Cmax of Ezetimibe Glucuronide (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Single Dose Administration of 400 mg Efavirenz) on Study Day 16
Description: as for outcome 16
Time Frame: study day 16
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 60.9 (29.5)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Cmax of Ezetimibe Glucuronide (Steady-state Pharmacokinetic After Chronic Treatment With 10 mg Ezetimibe and Concomitant Chronic Treatment With 400 mg Efavirenz) on Study Day 30
Description: as for outcome 16
Time Frame: study day 30
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Group
Number analyzed (Participants) | 12
ng/ml | 45.3 (14.6)
Statistical Analysis 1: Comparison: Study Group; Paired Wilcoxon-test between free ezetimibe with chronic treatment of efavirenz and free ezetimibe alone; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Group; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Study Group | Efavirenz Alone Single Dose | Ezetimibe Alone Multiple Dose | Ezetimibe Multiple Dose and Efavirenz Single Dose | Ezetimibe and Efavirenz Multiple Dose
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 8/12 | 3/12 | 7/12 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=12) | Efavirenz Alone Single Dose (N=12) | Ezetimibe Alone Multiple Dose (N=12) | Ezetimibe Multiple Dose and Efavirenz Single Dose (N=12) | Ezetimibe and Efavirenz Multiple Dose (N=12)
Belly ache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea NOS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache NOS (Nervous system disorders) | 5 (11) | 4 (4) | 3 (3) | 0 (0) | 3 (4)
Hot flushes (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (Nervous system disorders) | 10 (18) | 5 (5) | 0 (0) | 7 (7) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restlessness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No